CLINICAL TRIAL: NCT07128732
Title: The Effect of Peer Mentoring Training on Mentor Students' Life Skills: An Experimental Study
Brief Title: The Effect of Peer Mentoring Training on Mentor Students' Life Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Çağla Islattı Mutlu, Research Assistant, Nurse, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 09.2022.1529
Record Dates: First submitted 2025-07-28; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: Peer Mentoring; Life Skills
Keywords: Peer; mentoring; life skills; nursing student

STUDY DESIGN:
Intervention Model Description: There are two groups in the study: an experimental group that received peer mentoring training and a control group that received no training.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education (Experimental): Students in the education group will be given Peer Mentorship Training, which includes self-management and self-awareness, stress management, coaching and mentoring, critical thinking, problem-solving and decision-making, effective communication and relationship management. The training was conducted for 12 hours face-to-face and 3 hours online.
  Interventions: Other: Peer mentoring training
- Control (No Intervention): Students in the control group will not participate in the training.

INTERVENTIONS:
Other: Peer mentoring training — As part of the intervention, a 15-hour peer mentoring training program was implemented, covering topics such as self-management and self-awareness, stress management, coaching and mentoring, critical thinking, problem-solving and decision-making, effective communication and relationship management.
  Arms: Education

SUMMARY:
The aim of this study is to determine the impact of peer mentoring training on the life skills of mentored nursing students. The following hypothesis was investigated in the study:

H1: The life skills score of the intervention group that received peer mentoring training was higher than the life skills score of the control group that did not receive training.

As part of the study, the intervention group will receive peer mentoring training. Participants are required to attend at least half of the training program, which covers topics such as self-management and self-awareness, stress management, coaching and mentoring, critical thinking, problem-solving and decision-making, effective communication, and relationship management. The control group will not participate in the training.

Data were collected from participants for pretests and posttests before and after the training program.

DETAILED DESCRIPTION:
Mentoring, which is studied in diverse fields such as business, psychology, and health, also has various applications in education. Supporting the professional training and personal development of nursing students, enhancing academic success, and easing the process of settling into school or university are some of these applications. A mentor is an experienced person who helps and supports a mentee's learning. A mentee, on the other hand, is someone who receives career assistance and/or psychosocial support from a more senior and experienced mentor. Responsibilities of a mentor include support, information, protection, assigning responsibilities that will enable skill development, acting as a role model, counseling, ensuring the mentee's acceptance and acceptance of the institution, and friendship. Competence of mentors is crucial for a successful mentoring relationship.

Life skills are adaptable and positive behavioral skills that enable individuals to effectively cope with the demands, challenges, and obstacles of daily life. These skills support individuals for a productive life, help them adapt more easily to their situations, and are learnable skills. UNESCO (2008) defines life skills as: It defines life skills as psychosocial skills that can be learned and applied, such as self-awareness, problem-solving, critical thinking, and interpersonal skills. The World Health Organization (WHO), on the other hand, expands the definition of life skills, encompassing decision-making, problem-solving, coping with stress, coping with emotions, self-awareness, communication skills, creative thinking, empathy, and interpersonal skills.

This study was planned as a randomized controlled pretest-posttest experimental study to determine the effect of peer mentoring training on the life skills of mentor nursing students. The study was conducted between December 2022 and June 2023 at the Department of Nursing, Faculty of Health Sciences, of a state university. The study population consisted of third- and fourth-year students enrolled in the Department of Nursing, Faculty of Health Sciences, of a state university during the 2022-2023 academic year. The G*Power (v3.1.9.7) program was used to determine the sample size, and a total of 32 students were included, 16 in each group, taking into account possible losses. Before the study began, students were numbered and randomly assigned to either the experimental or control groups using a random number table. First, students were interviewed face-to-face to inform them about the study and invite them to participate. Informed consent was obtained from those who agreed to participate. For pre-test purposes, participants in the experimental and control groups were asked to fill out the Descriptive Information Form and the Life Skills Scale. Then, students in the experimental group received 15 hours of peer mentoring training. The training included presentations by faculty members specialized in self-management and self-awareness, stress management, coaching and mentoring, critical thinking, problem solving and decision-making, effective communication, and relationship management. Twelve hours of the training were conducted face-to-face. Due to the earthquake disaster in our country during the training period, education and training began to be conducted online. Therefore, three hours of the training were conducted online. The control group did not participate. After the training, students in the experimental and control groups were asked to complete the Life Skills Scale again for post-test purposes, and the final data were collected online. Ethics committee approval, institutional permission, and scale use permission were obtained before starting the research.

ELIGIBILITY:
Inclusion Criteria:

* Must be a third- or fourth-year student in the relevant department during the 2022-2023 academic year
* Students in the intervention group must be mentors in the peer mentoring program
* Attend at least half of the training sessions
* Participate in the research voluntarily
* Completely complete the data collection tool.

Exclusion Criteria:

* Being a first or second year student,
* Wanting to withdraw from the study for any reason,
* Filling out the data collection tool incompletely/incorrectly.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
Life skills scale scores | 6 months
  It is a five-point Likert-type scale consisting of 30 items and five sub-dimensions: coping with stress and emotions (7 items), empathy and self-awareness (7 items), decision-making and problem-solving (7 items), creative and critical thinking (5 items), and communication and interpersonal relationships (4 items). The scale does not contain negative statements. High scores indicate high life skills.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Ergün, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No